CLINICAL TRIAL: NCT00695110
Title: Phase II, Repeat Dose, Pharmacokinetic Study of Oral Testosterone Ester Formulations in Hypogonadal Men
Brief Title: Pharmacokinetic Study of Oral Testosterone (T) Ester Formulations in Hypogonadal Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clarus Therapeutics, Inc. (Industry)
Collaborators: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLAR-08005
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Results first posted 2021-06-24 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Hypogonadism
Keywords: testosterone; male hypogonadism; low testosterone
MeSH Terms: conditions — Hypogonadism; Eunuchism | interventions — testosterone undecanoate; testosterone enanthate; Food

STUDY DESIGN:
Intervention Model Description: All subjects were enrolled into a single group and proceeded through the four Treatment Periods 1-4 in a sequential manner.
Oversight: Data Monitoring Committee: No

ARMS (1):
- All study participants (Experimental): Treatment Period 1: Three capsules each containing 100 mg testosterone (T) as testosterone undecanoate (TU), twice daily (BID) for 7 days.
  Treatment Period 2: Two capsules each containing 200 mg T as TU and testosterone enanthate (TE), BID for 7 days.
  Treatment Period 3: Two capsules each containing 100 mg T as TU, BID for 8 days.
  Treatment Period 4: Two capsules each containing 150 mg T as TU and TE, BID for 7 days.
  Interventions: Drug: Oral testosterone undecanoate (TU) (300 mg T equivalents/dose); Drug: Oral testosterone undecanoate (TU) combined with testosterone enanthate (TE) (400 mg T equivalents/dose); Drug: Oral testosterone undecanoate (TU) (200 mg T equivalents/dose with and without food); Drug: Oral testosterone undecanoate (TU) combined with testosterone enanthate (TE) (300 mg T equivalents/dose)

INTERVENTIONS:
Drug: Oral testosterone undecanoate (TU) (300 mg T equivalents/dose) — Three capsules each containing 100 mg testosterone (T) as TU, BID. 300 mg T equivalents BID 30 minutes after initiation of breakfast and dinner meals for 7 days. A 7-14 day washout period occurred between successive Treatment Periods.
Drug: Oral testosterone undecanoate (TU) combined with testosterone enanthate (TE) (400 mg T equivalents/dose) — Two capsules each containing 100 mg T as TU and 100 mg T as TE, BID. 400 mg T equivalents BID 30 minutes after initiation of breakfast and dinner meals for 7 days. A 7-14 day washout period occurred between successive Treatment Periods.
Drug: Oral testosterone undecanoate (TU) (200 mg T equivalents/dose with and without food) — Two capsules each containing 100 mg T as TU, BID for 8 days. 200 mg T equivalents BID 30 minutes after initiation of meals (breakfast and dinner), except for Day 8 when the morning dose was administered fasting. A 7-14 day washout period occurred between successive Treatment Periods.
Drug: Oral testosterone undecanoate (TU) combined with testosterone enanthate (TE) (300 mg T equivalents/dose) — Two capsules each containing 150 mg T as TU and 150 mg T as TE, BID. 300 mg T equivalents BID 30 minutes after initiation of breakfast and dinner meals for 7 days.

SUMMARY:
The purpose of this pharmacokinetic study is to determine whether oral testosterone (T) ester formulations can be used effectively to treat men with low testosterone.

DETAILED DESCRIPTION:
Determination of the steady-state serum T pharmacokinetic profiles for two oral formulations of T-esters [testosterone undecanoate (TU) and TU combined with testosterone enanthate (TE)] administered bis in die (BID) to 29 hypogonadal adult male subjects. TU was evaluated in total daily doses of 400 and 600 mg equivalents of T given twice daily for 7 or 8 days; TU + TE was evaluated in total daily doses of 600 and 800 mg equivalents of T given twice daily for 7 days. All subjects were enrolled into a single group and proceeded through the four Treatment Periods 1-4 in a sequential manner. In Treatment Period 3 the effect of food on the study-state pharmacokinetics profile of the TU formulation was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male, ages 18-68
* Serum total T less than or equal to 275 ng/dL

Exclusion Criteria:

* Significant intercurrent disease of any type, in particular, liver, kidney or heart disease, uncontrolled diabetes mellitus or psychiatric illness.
* Abnormal prostate digital rectal examination, elevated prostate-specific antigen (PSA), American Urological Association (AUA) symptom score of >15, and/or history of prostate cancer.
* Hematocrit of <35 or >50%
* Body mass index (BMI) >36
* Serum transaminases > 2 times upper limit of normal or serum bilirubin > 2.0 mg/dL

Ages: 18 Years to 68 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald S Swerdloff, M.D., Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center; Gregory Flippo, M.D., Principal Investigator — Alabama Clinical Therapeutics, Inc.; Steven J. Kulback, M.D., Principal Investigator — Alabama Internal Medicine; Sherwyn Schwartz, M.D., Principal Investigator — dgd Research, Inc.
Locations (4):
- United States (4):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Alabama Internal Medicine, Birmingham, Alabama
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Los Angeles, California
  - dgd Research, Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yin AY, Htun M, Swerdloff RS, Diaz-Arjonilla M, Dudley RE, Faulkner S, Bross R, Leung A, Baravarian S, Hull L, Longstreth JA, Kulback S, Flippo G, Wang C. Reexamination of pharmacokinetics of oral testosterone undecanoate in hypogonadal men with a new self-emulsifying formulation. J Androl. 2012 Mar-Apr;33(2):190-201. doi: 10.2164/jandrol.111.013169. Epub 2011 Apr 7. PMID 21474786

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 45 subjects were screened at 4 study sites (1 university medical center and 3 clinical sites). 29 hypogonadal males met all eligibility requirements and were enrolled with first study drug administration on June 13, 2008.
Pre-assignment Details: After signing an informed consent form, subjects underwent a screening evaluation up to 28 days prior to the first dose of study drug. 29 subjects meeting the admission criteria, began Treatment Period 1 intervention (7 days) followed by a 7-14 day washout period and then proceeded to Treatment Periods 2-4. A 7-14 day washout period occurred between successive Treatment Periods. Treatment Periods 1, 2, and 4 had intervention for 7 days and Treatment Period 3 had intervention for 8 days.
Groups:
- All Study Participants: Repeat dose, single-group study including 4 treatment periods with a 7-14 day washout between successive periods:
  Treatment Period 1: Three capsules each containing 100 mg testosterone (T) as testosterone undecanoate (TU), BID, 30 minutes after initiation of breakfast and dinner meals for 7 days.
  Treatment Period 2: Two capsules each containing 200 mg T as TU and testosterone enanthate (TE), BID, 30 minutes after initiation of breakfast and dinner meals for 7 days.
  Treatment Period 3: Two capsules each containing 100 mg T as TU, BID for 8 days except for Day 8 when the morning dose was administered fasting.
  Treatment Period 4: Two capsules each containing 150 mg T as TU and TE, BID, 30 minutes after initiation of breakfast and dinner meals for 7 days.
Period: Treatment Period 1
Arm/Group | All Study Participants
Started | 29
Completed | 26
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Period: Treatment Period 2
Arm/Group | All Study Participants
Started | 26
Completed | 26
Not Completed | 0
Period: Treatment Period 3
Arm/Group | All Study Participants
Started | 26
Completed | 25
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Treatment Period 4
Arm/Group | All Study Participants
Started | 25
Completed | 24
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Data for all 29 subjects enrolled in this single group, four period study are included in the baseline measures at Treatment Period 1. No additional baseline measures were analyzed for successive Treatment Periods 2-4.
Groups:
- All Study Participants: Repeat dose, sequential cross-over study including 4 treatment periods with a 7-14 day washout between successive periods:
  Period 1: Three capsules each containing 100 mg testosterone (T) as testosterone undecanoate (TU), BID, 30 minutes after initiation of breakfast and dinner meals for 7 days.
  Period 2: Two capsules each containing 200 mg T as TU and testosterone enanthate (TE), BID, 30 minutes after initiation of breakfast and dinner meals for 7 days.
  Period 3: Two capsules each containing 100 mg T as TU, BID for 8 days except for Day 8 when the morning dose was administered fasting.
  Period 4: Two capsules each containing 150 mg T as TU and TE, BID, 30 minutes after initiation of breakfast and dinner meals for 7 days.
Arm/Group | All Study Participants
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Total Testosterone (ng/dL) [Mean (Standard Deviation); unit: ng/dL] | 169.0 (82.80)
Body Mass Index (BMI) (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 30.4 (3.43)
Height [Mean (Standard Deviation); unit: inches] | 69.9 (4.0)
Weight [Mean (Standard Deviation); unit: pounds] | 212.2 (38.68)

OUTCOME MEASURES:

1. Primary Outcome: Serum Testosterone Average Concentration (Cavg) (ng/dL)
Description: Sampling to determine serum T Cavg post AM and PM doses and for 24 hours in Treatment Periods 1, 2, and 4. Sampling to determine serum T Cavg post AM dose with food (Day 7) and fasting (Day 8) in Treatment Period 3.
Time Frame: 30 minutes pre-dose and 0, 1, 2, 4, 8, 12 hours and 0,1, 2, 4, 8, and 12 hours post respective AM/PM doses
Population: All available individual serum concentrations and pharmacokinetic parameter estimates were reported; missing data were not imputed. For 1 subject in Treatment Period 1 and 1 subject in Treatment Period 4 there were insufficient data to calculate all pharmacokinetic parameters.
Measure: Mean (Standard Deviation); unit: ng/dL
Groups:
- Treatment Period 1: Oral testosterone undecanoate (TU) (300 mg T equivalents/dose): Three capsules each containing 100 mg testosterone (T) as TU, BID, 30 minutes after initiation of breakfast and dinner meals for 7 days. A 7-14 day washout period occurred between successive Treatment Periods.
- Treatment Period 2: Oral testosterone undecanoate (TU) combined with testosterone enanthate (TE) (400 mg T equivalents/dose): Two capsules each containing 100 mg T as TU and 100 mg T as TE, BID. 400 mg T equivalents BID, 30 minutes after initiation of breakfast and dinner meals for 7 days. A 7-14 day washout period occurred between successive Treatment Periods.
- Treatment Period 3: Oral testosterone undecanoate (TU) (200 mg T equivalents/dose) with and without food): Two capsules each containing 100 mg T as TU, BID for 8 days 30 minutes after initiation of meals (breakfast and dinner), except for Day 8 when the morning dose was administered fasting. A 7-14 day washout period occurred between successive Treatment Periods.
- Treatment Period 4: Oral testosterone undecanoate (TU) combined with testosterone enanthate (TE) (300 mg T equivalents/dose): Two capsules each containing 150 mg T as TU and TE, BID, 30 minutes after initiation of breakfast and dinner meals for 7 days.
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4
Number analyzed (Participants) | 28 | 26 | 26 | 24
ng/dL
  Cavg (0-24): number analyzed (Participants) | 28 | 26 | 0 | 24
  Cavg (0-24) | 792 (254) | 654 (230) |  | 541 (289)
  Cavg (AM dose) with food | 765 (333) | 657 (294) | 518 (233) | 533 (385)
  Cavg (PM dose) with food: number analyzed (Participants) | 28 | 26 | 0 | 24
  Cavg (PM dose) with food | 819 (291) | 651 (236) |  | 548 (250)
  Cavg (AM dose) fasting: number analyzed (Participants) | 0 | 0 | 26 | 0
  Cavg (AM dose) fasting |  |  | 241 (106) |

2. Primary Outcome: Serum Testosterone Area Under Curve (AUC) (0-24) (ng•hr/dL)
Description: Sampling to determine serum T AUC post AM and PM doses and for 24 hours in Treatment Periods 1, 2, and 4. Sampling to determine serum T AUC with food (Day 7) and fasting (Day 8) in Treatment Period 3.
Time Frame: 30 minutes pre-dose and 0, 1, 2, 4, 8, 12 hours and 0,1, 2, 4, 8, and 12 hours post respective AM/PM doses
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (ng•hr/dL)
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4
Number analyzed (Participants) | 28 | 26 | 26 | 24
(ng•hr/dL)
  AUC (0-24): number analyzed (Participants) | 28 | 26 | 0 | 24
  AUC (0-24) | 19009 (6102) | 15693 (5527) |  | 12980 (6926)
  AUC (0-12) (AM dose) with food | 9179 (3990) | 7881 (3524) | 6217 (2792) | 6601 (4614)
  AUC (12-24) (PM dose) with food: number analyzed (Participants) | 28 | 26 | 0 | 24
  AUC (12-24) (PM dose) with food | 9830 (3489) | 7812 (2837) |  | 2894 (1267)
  AUC (0-12) (AM dose) fasting: number analyzed (Participants) | 0 | 0 | 26 | 0
  AUC (0-12) (AM dose) fasting |  |  | 2894 (1267) |

ADVERSE EVENTS:
Time Frame: Adverse Events, whether observed by the investigator, elicited during telephone contacts and/or study visits, reported in response to a query, or reported spontaneously by the subject were recorded from time of informed consent throughout Treatment Periods 1-4 (7-8 days/period) and all 7-14 day washout periods between treatment periods totaling approximately 100 days.
Groups:
- All Study Participants: Single group, repeat dose study including 4 treatment periods (7-8 days) and a 7-14 day washout between successive periods:
  Treatment Period 1: Three capsules each containing 100 mg testosterone (T) as testosterone undecanoate (TU), BID, 30 minutes after initiation of breakfast and dinner meals for 7 days.
  Treatment Period 2: Two capsules each containing 200 mg T as TU and testosterone enanthate (TE), BID, 30 minutes after initiation of breakfast and dinner meals for 7 days.
  Treatment Period 3: Two capsules each containing 100 mg T as TU, BID for 8 days except for Day 8 when the morning dose was administered fasting.
  Treatment Period 4: Two capsules each containing 150 mg T as TU and TE, BID, 30 minutes after initiation of breakfast and dinner meals for 7 days.
  The primary purpose of the study was to evaluate the pharmacokinetics of T following short-term, repeat-dose administration of various T doses in the form of TU or as a combination of TU + TE (7-8 days). Consequently, the AEs represent the integrated sum over all of the treatment groups in what was short-term T exposure compared to long-term efficacy and safety evaluations. Due to the short-term exposure to each intervention, changes in laboratory parameters were assessed at the end of the overall study and not the end of each treatment intervention.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 19/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=29)
Osteomyelitis (Infections and infestations) | 1 (1) — Osteomyelitis, right foot
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=29)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Elbow pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased AST and ALT (Investigations) | 1 (1)
Emesis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 7 (8)
Gastrointestinal reflux (Gastrointestinal disorders) | 2 (3)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hunger (General disorders) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2)
Viral herpes simplex (Infections and infestations) | 1 (1)
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea and vomiting (Gastrointestinal disorders) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. If the communication contains subject matter for which patent protection should be sought, the Sponsor will notify the PI whereupon the PI agrees to grant the Sponsor an additional 60 days to file documents necessary to protect such invention.